CLINICAL TRIAL: NCT06321757
Title: PREVAIL Paclitaxel-coated Balloon in Small Coronary Disease and High-bleeding Risk Patients
Acronym: PARIS
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC30-PARIS
Record Dates: First submitted 2024-02-16; First posted 2024-03-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
Keywords: drug-coated balloon; paclitaxel; small native vessel coronary artery disease; coronary stenoses
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with small native vessel coronary artery disease: - Patients with small native vessel coronary artery disease y/or patients with High Bleeding Risk
  Interventions: Device: Percutaneous Coronary Intervention with DCB and DAPT

INTERVENTIONS:
Device: Percutaneous Coronary Intervention with DCB and DAPT — * Patients with PCI (DCB) + standard DAPT standard dual antiplatelet therapy (DAPT)
  * Patients with PCI (DCB) + short DAPT

SUMMARY:
Post-market, prospective, observational, multicenter, non-intervention study, to demonstrate the effectiveness of drug-coated ballon (DCB)therapy in real-world patients with small native vessel coronary artery disease, and to demonstrate the safety of short dual antiplatelet therapy (7 days) in high-bleeding risk patients with native small vessel coronary artery disease treated with DCB therapy. A percutaneous coronary intervention (PCI) with DCB will be performed in patients with native vessel coronary artery disease based on the criterion of the treating physician.

DETAILED DESCRIPTION:
Post-market, prospective, multicenter, non-intervention study, to demonstrate the effectiveness of drug-coated ballon therapy in real-world patients with small native vessel coronary artery disease, and to demonstrate the safety of short dual antiplatelet therapy (7 days) in high-bleeding risk patients with native small vessel coronary artery disease treated with DCB therapy. A PCI with DCB will be performed in patients with native vessel coronary artery disease based on the criterion of the treating physician. The angiographic study will be analyzed in a core lab (icicorelab) blinded to the procedural outcomes and the patients' follow-up.

As per clinical practice, 1-year clinical follow-up of all the patients will be conducted with a first assessment at 30 days, a second assessment at 6 months, and one final assessment at 12 months.

Should the patient have an elevated bleeding risk -defined as concomitant therapy with oral anticoagulation or a PRECISE-DAPT score ≥ 25- patients will be included in a high-bleeding risk substudy. The antiplatelet therapy regime will be administered according to the local investigator and the treating medical team.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* PCI with DCB on native arteries with diameters < 3 mm.
* Indication for PCI in acute coronary syndrome or chronic coronary syndrome or silent angina with an indication for PCI.

syndrome or silent angina with an indication for PCI.

* If previous lesion preparation was required after which angiographic residual lesion should not exist with diameter stenosis > 30% or flow-limiting coronary dissections.
* All antithrombotic therapies administered prior to the procedure are accepted. Still, they can be changed after the procedure.
* Capacity to understand and sign the written informed consent.
* If the patient has a high-bleeding risk defined by 1) PRECISE-DAPT SCORE ≥ 25 or 2) an indication for concomitant oral anticoagulation he can be included in the high- bleeding risk substudy as long as he does not meet the specific exclusion criteria.

Exclusion Criteria:

Patients with:

* Concomitant lesions on vessels > 3 mm in diameter in the same coronary territory.
* PCI on in-stent restenoses.
* PCI on culprit lesions of acute coronary syndrome with ST segment elevation.
* Patients with an indication for PCI on additional non-culprit lesions of acute coronary syndrome with ST segment elevation may be included in the study, if only non-culprit lesions are considered for the study.
* Life expectancy <12 months
* Pregnancy.
* Participation in clinicaltrials.
* Inability to give the written informed consent.
* Specific exclusion criteria for the high-bleeding risk patient subgroup:
* Past medical history of stent thrombosis.
* Indication for dual antiplatelet therapy for a different reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: drug-coated ballon therapy in real-world patients with small native vessel coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 501 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of DCB therapy | 1 year
  Incidence of MACE, which is a composite endpoint including cardiac mortality, myocardial infarction, and new revascularization of the target lesion

SECONDARY OUTCOMES:
Cardiac death | 1 year
  Incidence of Cardiac death
All-cause mortality | 1 year
  Incidence of All-cause mortality
Target vessel myocardial infarction | 1 year
  Incidence of Target vessel myocardial infarction
New target lesion revascularization (TLR) | 1 year
  Incidence of New target lesion revascularization (TLR)
Target vessel failure (TVF) | 1 year
  Incidence of Target vessel failure (TVF)
Major bleeding | 1 year
  Bleeding defined as BARC (Bleeding Academic Research Consortium) criteria 2,3 or 5
Minor bleeding | 1 year
  Anemia, defined as Hb<12g/dL for women and <13g/dL for men
1-year MACE indicende (cardiac mortality, myocardial infarction, and new revascularization of the target lesion) in high-bleeding risk patients treated with a short dual antiplatelet treatment (7 days) | 1 year
  safety analysis of short DAP (dual antiplatelet therapy) in terms of thrombotic risk after PCI

CONTACTS AND LOCATIONS:
Locations (17):
- Portugal (2):
  - Ulslo-H.Santa Cruz, Carnaxide
  - ULS Santa Maria, Lisbon
- Spain (15):
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario de Cruces, Barakaldo
  - University Hospital HM Montepríncipe, Boadilla del Monte
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Clinico San Cecilio, Granada
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de Leon, León
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Kirtane AJ, Gupta A, Iyengar S, Moses JW, Leon MB, Applegate R, Brodie B, Hannan E, Harjai K, Jensen LO, Park SJ, Perry R, Racz M, Saia F, Tu JV, Waksman R, Lansky AJ, Mehran R, Stone GW. Safety and efficacy of drug-eluting and bare metal stents: comprehensive meta-analysis of randomized trials and observational studies. Circulation. 2009 Jun 30;119(25):3198-206. doi: 10.1161/CIRCULATIONAHA.108.826479. Epub 2009 Jun 15. PMID 19528338
- [Background] Kleber FX, Schulz A, Waliszewski M, Hauschild T, Bohm M, Dietz U, Cremers B, Scheller B, Clever YP. Local paclitaxel induces late lumen enlargement in coronary arteries after balloon angioplasty. Clin Res Cardiol. 2015 Mar;104(3):217-25. doi: 10.1007/s00392-014-0775-2. Epub 2014 Oct 28. PMID 25349065